CLINICAL TRIAL: NCT01477047
Title: Identification of Risk Factors of Prolonged Wound Healing Following Total Hip and Knee Arthroplasty
Brief Title: Identification of Risk Factors of Prolonged Wound Healing Following Primary Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirill Gromov, MD, PhD, Hvidovre University Hospital
Other Study IDs: 2011-41-6844
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Evaluate Surgical, Medical and Pharmacological Factors Influence on Wound Healing Following Primary Arthroplasty Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving primary hip or knee arthoplasty

SUMMARY:
Prolonged wound drainage following total joint replacement surgery has been shown to be a predictor of postoperative infection. Several factors have been associated with delayed wound healing and increased risk of infection. Namely hypertension, obesity, diabetes, smoking and autoimmune disease have been shown to have a detrimental effect on wound healing. The purpose of this study is to verify those findings and determine additional pharmacological, surgical and patient related factors that may result in prolonged wound drainage, prolonged hospital stay and increased risk of infection

DETAILED DESCRIPTION:
Study type: Prospective cohort study. Inclusion criteria: All patients receiving primary total hip or knee replacement surgery at Hvidovre Hospital from January 1st 2012 to December 31st 2014.

Exclusion criteria: none Intervention: none

New hypothesis to be tested:

1. Hypertension is associated with prolonged wound drainage and increased risk of infection
2. Patients receiving Statin treatment have decreased postoperative wound drainage and decreased risk of infection.
3. Patients receiving Bisphosphonate treatment have increased postoperative wound drainage and increased risk of infection.

Measured patient related risk variables: Age, sex, primary OA diagnosis, diabetes, smoking, BMI, alcohol consumption, autoimmune disease and hypertension will all be recorded upon admission of the patient to the hospital. Hypertension will be defined when a patient is diagnosed with HT previously to the surgery, receives medical treatment and have systolic / diastolic BP above 140/90 mmHg upon admission. Patients with normal BP upon admission receiving treatment for HT will be classified as having regulated HT. Patients with elevated BP upon admission without previous HT diagnosis will be classified as having newly diagnosed HT. "Smoking" will de divided into smokers, non-smokers and former smokers. Further on, average number of cigarettes pr day during the last month will be recorded for current smokers.

Measured pharmacological risk variables: Use of statins, bisphosphonates, anticoagulants, NSAID's and corticosteroids on time of admission will be recorded.

Measured surgical risk variables: Surgery time, pneumatic tourniquet time, peroperative blood loss, postoperative decrease in hemoglobin levels, surgical complications, antibiotic and bleeding prophylaxis will be recorded by the surgeon upon completion of the surgery.

Outcome measures: Wound-oozing time, length of hospital stay, wound infections, and surgical revision. Wound will be defined as actively draining if the gauze covering the wound is wet to the edges or if fluid is noted to be originating from the surgical site. The nursing staff will record wound drainage during the hospital stay and the patient will be instructed in self-assessment upon dismissal using patient-diary. Wound drainage will be recorded twice a day: before- and afternoon. All patients are seen in outpatient clinic for staple removal and control of the self -assessment drainage-diary 3 weeks after surgery. Time when the wound appeared dry will be noted. Presence or absence of clinical infection will be noted according to ASEPSIS criteria.

Statistical analysis: Multiple linear regression analysis will be performed to model the effects of the measured risk variables on the time to a dry wound, length of hospital stay and risk of wound infection.

Data collection: All data collection will be anonymous. Patient consent is not required since the study involves evaluation of existing data and records and individual subjects can not be identified either directly or through identifiers linked to the subject. The data collection will be reported to "Datatilsynet".

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving primary hip or knee arthroplasty at Hvidovre Hospital from january 2012 to january 2014.

Exclusion Criteria:

* Not willing to participate.
* Drop out at 3 week follow up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving primary hip or knee arthroplasty at Hvidovre Hospital from january 2012 to january 2014.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Wound drainage time | 3 weeks

SECONDARY OUTCOMES:
Clinical infection | months

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark